CLINICAL TRIAL: NCT03684200
Title: Hip Adductor Muscle Strength Changes With the Copenhagen Adductor Exercise in Male Football (Soccer) Players.
Brief Title: The Copenhagen Adductor Exercise Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Mr Jack Dawkins, Principal Investigator, University of Bath
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UBath
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Eccentric Hip Adduction Strength

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Copenhagen adductor exercise (Experimental): 20 players allocated to the Copenhagen adductor exercise group complete a progressive strengthening programme comprising of the Copenhagen adductor exercise over a period of 6 weeks. They will complete two exercise sessions a week consisting of one set of the Copenhagen adductor exercise. The exercise will be performed on each side. The training load will increase from 5 repetitions in week 1, to 15 repetitions in week 6. The exercise programme is performed at the end of the warm-up of a regular football training session.
  Interventions: Other: Copenhagen adductor exercise
- Control (No Intervention): 19 players allocated to the control group will be asked not to perform the Copenhagen adductor exercise or any other specific strength training for the adductor muscles and to continue to play football as usual.

INTERVENTIONS:
Other: Copenhagen adductor exercise — The active player is supported on one forearm on the floor and the upper arm is resting along their side. The supporting partner places their hands at the ankle and the knee of the upper leg. The active partner raises their body from the floor and adducts both legs in a three second movement until the body reaches a straight line. The body is then lowered to the ground in a three second movement, the foot of the lower leg touches the ground before performing another repetition.
  Other Names: Adductor bridge exercise
  Arms: Copenhagen adductor exercise

SUMMARY:
The purpose of this study is to investigate the efficacy of a 6-week intervention, using the Copenhagen adductor exercise, on adductor muscle strength in sub-elite male footballers. Secondly, it will also examine the effect of a 3-week detraining period, after stopping the Copenhagen adductor exercise, on adductor muscle strength.

The primary outcome measure is eccentric hip adduction strength measured using a handheld dynamometer. Additionally, peak isometric adductor squeeze strength will also be measured using a handheld dynamometer.

The hypothesis is that strength training of the adductor muscles elicited by the Copenhagen adductor exercise will result in enhanced eccentric hip adduction strength.

ELIGIBILITY:
Inclusion Criteria:

* Sub-elite English football player
* Age 18-26
* Participant can read, speak and understand English.
* Participant can receive and reply to texts on a cell phone using Short Message Services (SMS).
* Able to participate fully in competitive football training at time of testing.

Exclusion Criteria:

* Hip and groin pain resulting in loss of football training and matches in the 2 months prior to commencement of the trial.
* Specific strength training of the adductor muscles (>/1 week) in the 2 months prior to commencement of the trial.
* Participant cannot attend strength testing sessions during the study.

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Eccentric hip adduction strength measured using a handheld dynamometer | Measured after intervention period (at week 6)
  Lafayette handheld dynamometer (model: 01165) will be used to produce force values in Newtons.

SECONDARY OUTCOMES:
Eccentric hip adduction strength measured using a handheld dynamometer | Measured during intervention period (at week 3)
  Lafayette handheld dynamometer (model: 01165) will be used to produce force values in Newtons.
Eccentric hip adduction strength measured using a handheld dynamometer | Measured prior to and after intervention period (at week 0, 7, 8 and 9)
  Lafayette handheld dynamometer (model: 01165) will be used to produce force values in Newtons.
Peak isometric adductor squeeze strength measured using a handheld dynamometer | Measured after intervention period (at week 6)
  Lafayette handheld dynamometer (model: 01165) will be used to produce force values in Newtons.
Peak isometric adductor squeeze strength measured using a handheld dynamometer | Measured during intervention period (at week 3)
  Lafayette handheld dynamometer (model: 01165) will be used to produce force values in Newtons.
Peak isometric adductor squeeze strength measured using a handheld dynamometer | Measured prior to and after intervention period (at week 0, 7, 8 and 9)
  Lafayette handheld dynamometer (model: 01165) will be used to produce force values in Newtons.
Maximal weekly delayed onset of muscle soreness (DOMS) | Measured during intervention period (at week 1, 2, 3, 4, 5 and 6)
  Measured using a 0-10 numeric rating scale (NRS).
Rate of perceived exertion (RPE) at each session training session. | Measured during intervention period (at week 1, 2, 3, 4, 5 and 6)
  Measured using the 6-20 Borg Rating of Perceived Exertion Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Physio & Sports Science Centre, University of Bath, Bath, Avon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided